CLINICAL TRIAL: NCT00293553
Title: Clinical Approaches to Ileal Pouch Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R03 DK67275 (completed 2007); R03DK067275 (NIH)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis

INTERVENTIONS:
Procedure: Electronic Barostat

SUMMARY:
Total proctocolectomy and ileal pouch-anal anastomosis is the surgical treatment of choice for patients with medically refractory ulcerative colitis, ulcerative colitis with dysplasia or cancer, and patients with familial adenomatous polyposis. Pouchitis, an inflammatory process of the ileal pouch, is the most common long-term complication. Increased stool frequency, abdominal pain, and pelvic discomfort are suggestive of pouchitis, approximately 40% of patients with these symptoms have no or minimal inflammation of the pouch or rectal cuff on endoscopy and histopathology. These patients have a condition resembling irritable bowel syndrome (IBS), which we termed the irritable pouch syndrome (IPS). The RATIONALE and FEASIBILITY for the proposed study are: 1) IPS occurs in a substantial number of patients with IPAA, significantly affecting the quality of life. However, IPS is rare in the general population, and is considered an orphan disease. Studies such as those we propose can only be conducted in centers with a large number of patients with IPAA. The Cleveland Clinic has maintained the world's largest ileal pouch registry, with a total of more the 2,500 patients; 2) a series of investigations on the diagnosis and treatment of patients with inflammatory or functional diseases of IPS, notably the initial study of IPS, have been conducted by our team; 3) In contrast to IBS, the pathophysiology and treatment of IPS have not been studied. Our HYPOTHESES are that 1) similar to IBS, visceral hypersensitivity may play a role in the pathogenesis of IPS, and 2) amitriptyline, a safe and effective agent for patients with IBS, will be more effective than placebo in alleviating symptoms and improving quality of life in patients with IPS. The AIMS of the study are to 1) investigate visceral hypersensitivity using barostat examination of the pouch; 2) conduct a randomized, placebo-controlled clinical trial evaluating the use of amitriptyline in IPS.

ELIGIBILITY:
Inclusion Criteria:(must meet ALL of the following criteria);

* Having a history of UC and more than 1 year from TPC/IPAA
* Meet diagnostic criteria of IPS, i.e.
* Symptoms of diarrhea and abdominal pain, with PDAI symptoms score > (range 2-6).
* Duration of symptoms > 12 weeks in the preceding 12-months period
* Pouch endoscopy shows no evidence of inflammation of the ileal pouch and rectal cuff
* No antibiotic therapy, aspirin, or non-steriodal anti-inflammatory drugs for 2 weeks prior to entry into the study; no antidepressant and or anti-anxiety medicines for at least 4 weeks.

Exclusion Criteria:(may meet ANY of the following criteria);

* A history of development of side effects from amitriptyline
* IPAA for FAP; celiac disease; chronic pouchitis; Crohn's disease; pouch stricture or anastomotic leak
* Urinary retention, glaucoma, use of MAO inhibitors within past 14 days; acute recovery phase following myocardial infarction; pregnancy
* Psychiatric disorder, including major depression, which requires medical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Shen, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States